CLINICAL TRIAL: NCT03341806
Title: Phase I Study of PD-L1 Inhibition With Avelumab and Laser Interstitial Thermal Therapy in Patients With Recurrent Glioblastoma
Brief Title: Avelumab With Laser Interstitial Therapy for Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Adilia Hormigo, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-1866
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Glioblastoma; GBM
Keywords: GBM; LITT; Laser Interstitial Thermal Therapy; Bavencio; immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Recurrent Glioblastoma (Experimental): Part A - Avelumab Part B - Avelumab + MRI-guided LITT therapy
  Interventions: Drug: Avelumab; Combination Product: MRI-guided LITT therapy

INTERVENTIONS:
Drug: Avelumab — Avelumab will be administered intravenously every 2 weeks at a dose of 10 mg/kg for 2 cycles
Combination Product: MRI-guided LITT therapy — (Part B) prior to receiving Avelumab 10 mg/kg every 2 weeks + LITT

SUMMARY:
The purpose of the study is to characterize the safety and tolerability of avelumab in combination with Laser Interstitial Thermal Therapy (LITT) for blood barrier disruption in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
This is an open label, non-randomized Phase I study of intravenous avelumab every 2 weeks to be administered after real-time MRI-guided LITT therapy for patients with a first recurrence of a glioblastoma.

The primary objective of the study is to characterize the tolerability and safety profile of avelumab in combination with MRI guided LITT administered to patients diagnosed with recurrent GBM.

Part A, the initial cohort of patients will be treated with intravenous avelumab alone. Part B, patients will receive avelumab in combination with MRI-guided LITT to characterize the tolerability and safety of the combined treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven GBM from the initial resection.
* Patients must have a life expectancy > 16 weeks. Patients must have a Karnofsky performance status of ≥ 60 or ECOG 0 - 2
* Patient's requirement for dexamethasone should be ≤ 4mg daily or a stable dose at enrollment.
* Patients must have adequate bone marrow, hepatic and renal function and hemoglobin and the test musts be performed within 14 days prior to study Day 1.
* Highly effective contraception for both male and female subjects if the risk of conception exists.

Exclusion Criteria:

* Known history of autoimmune disorder except diabetes mellitus type 1, vitiligo or hypothyroidism only requiring hormone replacement
* Patients who have received any other therapeutic investigational agent within 30 days of enrollment with the exception of the personalized MTA vaccine (NCT03223103) that can be continued throughout the study.
* Patients who have received any other therapeutic investigational agent within 30 days of enrollment or prior
* Prior placement of intracavitary BCNU-impregnated wafers (Gliadel).
* Prior treatment with checkpoint inhibitors, CTL-4 antibody or other immunotherapy agents
* Presence of any other active malignancy or prior history of malignancy, except for: basal cell carcinoma of the skin, cervical carcinoma in situ, early stage prostate carcinoma not requiring active treatment.
* Prior organ transplantation, including allogeneic stem cell transplantation
* Significant acute or chronic infections including, among others: HIV, AIDS, HBV
* Pregnancy or lactation

Contact site for full inclusion/exclusion list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity level | 4 weeks
  Toxicity will be measured by severity of Adverse events with toxicity grading defined by Cancer Therapy Evaluation Program's (CTEP) v4.0 of National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) scale.
Objective response rate (ORR) | 6 months
  Tumor response to treatment with avelumab in combination with MRI-guided LITT administered to patients with recurrent GBM by estimation of the objective response rate (ORR) -classified according to the RANO Response Criteria (Proportion of Complete Response, Partial Response, Stable Disease and Progressive Disease)

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  The % of progression free survival at 6 months
Overall response rate | 6 months
  Overall response rate (proportion of partial and complete responses) will be evaluated according to Rano criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Adilia Hormigo, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No